CLINICAL TRIAL: NCT02225678
Title: Feasibility of Using an Eosinophil-Specific Biomarker-(Eosinophil Peroxidase) in Clinical Practice
Brief Title: Minimally Invasive Biomarker for Asthma Disease Severity
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James J. Lee, Ph.D., PI, Mayo Clinic
Other Study IDs: 14-001168
Record Dates: First submitted 2014-07-24; First posted 2014-08-26 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Asthma; Healthy
Keywords: healthy volunteers; asthma; sputum eosinophils
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum
Oversight: Data Monitoring Committee: No

SUMMARY:
Can a clinical test be developed that could help manage asthma symptoms?

DETAILED DESCRIPTION:
Project goals:

Develop a point-of-service assay to assess eosinophilic airway inflammation

Proposal Specific Aims:

1. To establish the infrastructure and test the feasibility of sputum collection in a clinical setting as a minimally invasive patient sampling process for biomarker testing
2. To transform the laboratory-based eosinophil peroxidase (EPX) ELISA detection assay into a clinic-friendly assessment that does not require sophisticated laboratory equipment

ELIGIBILITY:
Asthma subjects:

Inclusion

* Provider diagnosed asthma
* FeNO>50 ppb
* FEV1 > 1.0 Liter

Exclusion

* COPD by history
* Bronchiectasis by history
* Pregnant participants

Normal subjects:

Inclusion

- Age matched to asthma subjects

Exclusion

* Any eosinophil disorder by history
* Asthma by history
* Rhinitis or sinusitis by history

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asthma patients healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Sputum Induction | 10 minutes
  Primary Outcome measure via EPX levels (at point of care) in the sputum of asthma patients and control subjects as a means of demonstrating the ability to use this biomarker approach in a clinical setting.

CONTACTS AND LOCATIONS:
Overall Officials: James Lee, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States